CLINICAL TRIAL: NCT01143129
Title: Postoperative New-onset Atrial Fibrillation in Cardiac Surgery: An Explanatory Study of the Prophylactic Effect of Corticosteroids (DECS-PNAF Project)
Brief Title: Postoperative New-onset Atrial Fibrillation in Cardiac Surgery: DECS-PNAF Project
Acronym: DECS-PNAF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, J.M. Dieleman, Anesthesiologist in training, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DECS-PNAF
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-02

CONDITIONS: Atrial Fibrillation; Cardiac Surgery
Keywords: Atrial fibrillation; Cardiac surgery; Cardiopulmonary bypass; New-onset
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dexamethasone (Experimental): Single dose of dexamethasone (1 mg/kg) at the start of the cardiac surgical procedure
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone — Single dose (1 mg/kg) at start of cardiac surgical procedure
  Arms: dexamethasone
Drug: Placebo — Placebo solution in a comparable amount to the experimental drug (0.05 mL/kg)
  Arms: Placebo

SUMMARY:
The DExamethasone for Cardiac Surgery - Postoperative New-onset Atrial Fibrillation (DECS-PNAF) project described in this protocol aims to elucidate how corticosteroids protect cardiac surgical patients from Postoperative New-onset Atrial Fibrillation (PNAF). Patients will be randomized to receive either a single high dose of dexamethasone or a placebo. Continuous ECG-monitoring, echocardiography and biochemical and genomic analyses will be used to investigate the mechanisms responsible for the known protective effect of corticosteroids in the development of PNAF.

DETAILED DESCRIPTION:
Postoperative new-onset atrial fibrillation (PNAF) is a common complication after cardiac surgery, affecting up to 60% of patients. PNAF has been associated with a higher incidence of adverse postoperative outcomes including long-term mortality, and leads to an increased use of resources and higher social costs.

Many studies have investigated potential determinants of PNAF. Established determinants can grossly be divided into inflammatory factors, cardiac functional (echographic) parameters, cardiac electrophysiologic properties and other (demographic) risk factors. Also, a substantial number of studies have investigated pharmacological prophylactic strategies. In these studies, the highest effectiveness has been shown for strategies involving either betablockers, statins and, more recently, corticosteroids.

The DExamethasone for Cardiac Surgery - Postoperative New-onset Atrial Fibrillation (DECS-PNAF) project described in this protocol aims to elucidate how corticosteroids protect cardiac surgical patients from PNAF. The modulating effect of intraoperative prophylactic high-dose dexamethasone administration on the categories of perioperative determinants of PNAF mentioned above will be studied in 164 coronary artery bypass grafting surgery patients. For this, multiple perioperative assessments will be performed using, for example, repeated biochemical assessment of inflammation, genomic analysis of (mainly inflammatory) single nucleotide polymorphisms, continuous electrocardiographic (Holter) monitoring and transesophageal echocardiography.

The DECS-PNAF project is one of the first prospective studies to combine a detailed assessment of multiple categories of PNAF determinants. Moreover, it is unique in studying the effect of prophylactic corticosteroid administration on every one of these determinants.

ELIGIBILITY:
Inclusion Criteria:

* On-pump coronary artery bypass graft (CABG)

Exclusion Criteria:

* age < 18 years
* preexisting cardiac rhythm disturbances

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-01; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Atrial fibrillation | 5 days (postoperatively)

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands